CLINICAL TRIAL: NCT05072132
Title: Returning Genetic Results on Arsenic Susceptibility to Bangladeshi Research Participants
Brief Title: Returning Genetic Results on Arsenic Susceptibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB20-1058
Record Dates: First submitted 2021-09-15; First posted 2021-10-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Arsenic Exposure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inefficient metabolizers (Experimental): Participants will be selected based on being inefficient arsenic metabolizers. A standard informational intervention will be provided, reminding them of the effects of arsenic exposure and strategies to reduce their exposure. This intervention group will additionally be provided information on their arsenic metabolism efficiency (i.e., their genetic results indicating they are inefficient metabolizers and at increased risk for arsenic toxicities).
  Interventions: Other: Personal information on genetic susceptibility to arsenic toxicity; Other: standard information on arsenic exposure reduction
- Efficient metabolizers (Experimental): Participants will be selected based on being efficient arsenic metabolizers. A standard informational intervention will be provided, reminding them of the effects of arsenic exposure and strategies to reduce their exposure. This intervention group will additionally be provided information on their arsenic metabolism efficiency (i.e., their genetic results indicating they are efficient metabolizers and at decreased risk for arsenic toxicities).
  Interventions: Other: Personal information on genetic susceptibility to arsenic toxicity; Other: standard information on arsenic exposure reduction
- Control group (Active Comparator): The control group will consist of a random sample of HEALS participants. A standard informational intervention will be provided, reminding them of the effects of arsenic exposure and strategies to reduce their exposure. No information on arsenic metabolism efficiency will be provided during the study period (option to receive after the study)
  Interventions: Other: standard information on arsenic exposure reduction

INTERVENTIONS:
Other: Personal information on genetic susceptibility to arsenic toxicity — The intervention groups will receive information regarding their genetic results that informs them of their arsenic metabolism efficiency. They will receive this information through a factsheet appropriate for a lay audience. The factsheet will contain information regarding arsenic metabolism and its role in removing arsenic from the body. The factsheet will describe how there is variability among individuals with respect to the efficiency with which arsenic is removed from the body, due to inherited differences in genes that affect arsenic metabolism. The factsheet describe how slower metabolizers remove arsenic slower from the body, which leads to increased in toxicity risk. The factsheet will inform participants in the intervention groups that they have been identified as a slow/fast metabolizer of arsenic based on their genes. This information will be given to participants by the URB staff, with a study physician available to address questions and concerns from the participant.
  Arms: Efficient metabolizers; Inefficient metabolizers
Other: standard information on arsenic exposure reduction — In this study, intervention and control groups will receive a standard informational intervention which will remind them of the effects of arsenic exposure and potential strategies that can be implemented to reduce their exposure.

SUMMARY:
In recent years, returning genetic results to research participants has become a topic of debate, with a growing consensus that researchers should offer to return incidental findings and research results to participants. Currently, the research and debates surrounding return of results (ROR) have primarily taken place in high-income countries. Less attention has been paid to ROR in lower-resource countries. However, research participants in these settings may have additional threats, barriers, and/or competing interests that reduce the benefit or relevance of receiving genetic results.

Arsenic is a toxic metal. Exposure to arsenic increases a person's risk for cancer, especially in the lung, kidney, bladder and skin. Many people in Bangladesh are exposed to elevated environmental levels of arsenic through naturally contaminated drinking water. People who metabolize arsenic (remove it from their body) slower compared to people who metabolize arsenic more efficiently are at higher risk for arsenic toxicities (e.g. cancer).

The investigators have designed a study in which they plan to enroll individuals who have had consistently high urine As levels (≥200 µg/g creatinine) based on 15-20 years of follow-up data. The treatment and control groups will be selected based on genotype (i.e. inefficient and efficient As metabolizers, respectively), allowing for the selection of the groups to be quasi-random (based on inherited genotypes). A standard informational intervention will be provided to both the treatment and controls groups, reminding them of the effects of As exposure and strategies to reduce their exposure.

The research question is whether the treatment group will, have a larger decrease in urine arsenic levels compared to the control group, indicating that the ROR intervention caused a change in water-seeking behavior leading to lower arsenic exposure.

DETAILED DESCRIPTION:
Abstract: In recent years, returning genetic results to research participants has become a topic of debate, with a growing consensus that researchers should offer to return incidental findings and research results to participants. The research and debates surrounding return of results (ROR) have primarily taken place in high-income countries. Less attention has been paid to ROR in lower-resource countries. The investigators propose to examine the impact of ROR on behavioral changes related to arsenic exposure reduction within The Health Effects of Arsenic Longitudinal Study (HEALS) cohort (IRB18-1331). This cohort study is located in Araihazar, Bangladesh, a rural area of Bangladesh with substantial exposure to arsenic through naturally contaminated drinking water from local wells. In this cohort, the investigators have participant data on inherited genetic variation known to impact arsenic metabolism efficiency and risk for arsenic toxicities. These genetic data allow us to identify participants who are inefficient (vs. efficient) arsenic metabolizers. The investigators previously surveyed 200 HEALS participants regarding their attitudes towards receiving information about their genetic susceptibility to arsenic toxicity, and 100% of the participants indicated they wanted to receive this information. The investigators are proposing a study in which they enroll adults who have had consistently high urine arsenic levels (≥200 µg/g creatinine) based on 15-20 years of follow-up data. The 2 intervention groups (n=200) will be selected based on genotype (i.e. inefficient and efficient arsenic metabolizers, respectively), allowing for the selection of the groups to be quasi-random (based on inherited genotypes). The control group (n=100), will be selected at random within the HEALS participants who have had consistently high urine arsenic levels. The intervention will consist of three arms: 2 intervention groups (n=200) and 1 control group (n=100). The intervention arm will consist of two groups; intervention 1 and intervention 2. Participants in intervention 1 group will be selected based on being inefficient arsenic metabolizers, while participants in intervention 2 group will be selected based on being efficient arsenic metabolizers. The control group will consist of a random sample of HEALS participants. A standard informational intervention will be provided to both the intervention and controls groups, reminding them of the effects of arsenic exposure and strategies to reduce their exposure. The intervention groups will additionally be offered information on their arsenic metabolism efficiency (i.e., their genetic results indicating they are inefficient/efficient metabolizers and at increased/decreased risk for arsenic toxicities). Six months after the intervention, the urine arsenic levels of all groups will be measured. The investigators hypothesize that the intervention 1 group (inefficient arsenic metabolizers) will have a larger decrease in urine arsenic levels compared to the control group. The investigatorshypothesize that the intervention 2 group will have urine arsenic levels that differ from intervention 1 group

Specific Aims:

Aim 1. To enroll arsenic-exposed individuals to an intervention study to assess the impact of returning information on genetic susceptibility on arsenic exposure levels. To achieve this aim, The investigators will first recruit HEALS participants (residing in Araihazar, Bangladesh) with consistently high arsenic exposure (based on >15 years of exposure data). Using genetic information to perform quasi-randomization, the investigators will then assign low-efficiency metabolizers to the intervention 1 arm and high-efficiency metabolizers to the intervention 2 arm(return of genetic results + exposure reduction information) and the control arm (exposure reduction information only).

Aim 2. To assess the impact of the ROR intervention on arsenic exposure levels, the investigators will collect urine samples 6 months after the intervention and compare the arsenic levels to arsenic levels assessed in urine at baseline. The investigators will test the association between the intervention arms and the change in arsenic levels between baseline and follow-up.

Background Returning genetic results to research participants has become a topic of debate in recent years due in part to increasing availability of whole-genome genotyping and sequencing data and an improved understanding of genetic causes of disease. Whole genome sequencing data can contain information relevant to the health care of a research participant, although not necessarily relevant to the research questions; this has been termed "incidental findings." There is a growing consensus that researchers should offer to return such incidental findings to research participants. Groups such as the American College of Medical Genetics (ACMG) have provide recommendations regarding which genes and variants should be considered "medically relevant and offered to participants as part of the incidental findings. There is also a trend among researchers and funders to make research participants' genetic data freely available to them should participants want to access to it. These types of data could be specific research results (i.e., the specific genetic variants[s] under study in meeting a research project's aims) or genome-wide measures of genetic variation (potentially communicated as polygenic estimates of risk for specific disease or as an interpretation of participants' genetic ancestry). It has been suggested that providing participants their genetic results is one way by which researchers can demonstrate respect for participants and enhance participants' engagement in research.

Study overview This study's primary goals are to test the feasibility and benefits of returning genetic results to a population in a rural and low resource setting. To accomplish the specific aims, the investigators will use data from the HEALS cohort from which they have previously obtained information regarding arsenic exposure as well as genomic information from Bangladeshi adults (age 18-70). Participants within this cohort will be eligible for this intervention study if they have had consistently high urine arsenic levels throughout the follow-up period (15-20 years of information). The information and knowledge gained from this study is critical for advancing understanding the potential benefits of returning genetic results within a low resource setting.

The investigators will collaborate with UChicago Research Bangladesh (URB) to enroll individuals from the HEALS cohort in Araihazar, Bangaldesh. URB will identify HEALS participants who have had consistently high urine arsenic levels (≥200 µg/g creatinine) based on 15-20 years of follow-up data. Intervention1 and intervention 2 groups will be selected based on genotype (i.e. inefficient and efficient arsenic metabolizers, respectively), allowing for the selection of the groups to be quasi-random (based on inherited genotypes). The control group will be selected randomly from HEALS participants. At initial contact (Time 1), URB filed staff in Araihazar will obtain urine samples from all participants. A standard informational intervention will be provided to intervention and controls groups, reminding them of the effects of arsenic exposure and strategies to reduce their exposure. The intervention groups will additionally be offered information on metabolism efficiency (i.e., their genetic results). Six months after the onset of the intervention (Time 2), the urine arsenic levels of both intervention and control groups will be measured again.

Duration The length of the data collection period for each participant will be 6 months. The initialization of the study will be Time 1, at which the first urine sample will be obtained, 6 months later (Time 2) the URB researchers will follow-up with the participants to obtain the last urine sample for this study. Given that data collection will be staggered across participants, collection of all urine samples is expected to take 1 year. Measurement of arsenic in those samples will take 6 months, and downstream analyses of data will take another 6 months. So the investigators expect ~2 years for this study once data collection has begun.

Location Collection of biospecimens and questionnaire data will take place in Araihazar, Bangladesh. The URB has local offices in this area. Arsenic measurement will occur at the University of Illinois in Chicago. Data analyses will occur at the University of Chicago.

Methodology:

Study population and participant selection: All participants will be recruited from the Health Effects of Arsenic Longitudinal Study (HEALS) in Araihazar, Bangladesh, a study that has >20,000 participants. HEALS is a prospective study of health outcomes associated with arsenic exposure through drinking water in a cohort of adults in Araihazar, Bangladesh, a rural area east of the capital city, Dhaka. Trained study physician conducted in-person interviews, clinical evaluations (including ascertainment of skin lesions), and urine collection at baseline and follow-up visits (every 2 years). Blood samples were also collected from the participants at baseline.

Type and number of experimental subjects: For this present study, Uchicago Research Bangladesh (URB) study staff will work to identify patients who meet the inclusion and exclusion criteria from the established HEALS cohort study during which the URB staff will obtain informed consent. The inclusion criteria for the study are HEALS cohort members (age 18-70) who have had consistently high urine arsenic levels (≥ 200 µg/g creatinine) based on 15-20 years of follow-up data and participants who have genetic information regarding the AS3MT variant that classifies them as being an inefficient or efficient arsenic metabolizer. The exclusion criteria for this study would be HEALS members who are missing baseline urine samples as well as those who are missing the latest follow-up urine samples. There will be a total of 300 subjects enrolled,100 for the intervention 1 group, 100 for the intervention 2 group and 100 for the control group. The investigators will collect urine samples from each participant to assess current levels of arsenic exposure. Urine samples will be shipped to the University of Chicago. Information regarding each HEALS participant's well usage will be updated at baseline.

Genetic information and Classification of slow vs. Fast metabolizers: Once consumed, inorganic arsenic is converted to mono- and di-methylated (DMA) forms. DMA, expressed as a percentage of urinary arsenic, is a measure of arsenic metabolism efficiency (AME). Common variation in the 10q24.32 region, containing the arsenic methyltransferase (AS3MT) gene, is associated with AME. Additionally, a genetic variant in the formiminotransferse cyclodeaminase (FTCD) gene is associated with AME. FTCD is critical for catabolism of histidine, a process that generates one-carbon units that can enter the one-carbon/folate cycle, which provides methyl groups for arsenic metabolism. In the HEALS cohort, these genetic variants in FTCD and AS3MT together explain ~10% of the variation in DMA% and have clear effects on risk for arsenic toxicity (i.e. arsenic-induced skin lesions). These inherited genetic variants will be used in the present study to classify participants as efficient or inefficient arsenic metabolizers.

Intervention (receiving information on arsenic): In this study, intervention and control groups will receive a standard informational intervention which will remind them of the effects of arsenic exposure and potential strategies that can be implemented to reduce their exposure. In addition, the intervention groups will receive information regarding their genetic results that informs them of their arsenic metabolism efficiency. The intervention groups will receive this information through a factsheet appropriate for a lay audience. The factsheet will contain information regarding arsenic metabolism and its role in removing arsenic from the body. The factsheet will describe how there is variability among individuals with respect to the efficiency with which arsenic is removed from the body, due to inherited differences in genes that affect arsenic metabolism. The factsheet will connect metabolism speed with toxicity risk. In other words, slower metabolizers remove arsenic slower from the body compared to others while fast metabolizers remove arsenic faster from the body compared to others. This leads to increased risk for arsenic toxicities, normal arsenic metabolizer remove arsenic from the body at an average rate, and fast arsenic metabolizers remove arsenic from the body faster than most other people, which leads to decreased toxicity risk. Lastly, the factsheet will inform the participants in the intervention groups that they have been identified as a slow/fast metabolizer of arsenic based on their genes. This information will be given to participants by URB staff, with a study physician available during the study visit who would be able to address additional questions and concerns from the participant. The control group will not receive the information regarding their genetic results that informs them of their arsenic metabolism efficiency.

Arsenic Assessment and Urine Sample: Urine samples will be obtained by URB study staff at Time1 (initial contact) and Time2 (Six months after the onset of the intervention). The investigators plan to assess arsenic exposure from urine samples from all recruited participants. Prior studies have demonstrated high correlation between water arsenic levels and urinary arsenic. Urine arsenic will be measured using Inductively Coupled Plasma Mass spectrometry (ICPMS) at the CACHET (The Chicago Center for Health and Environment) biomarkers core facility at UIC (University of Illinois at Chicago).

Questionnaires: All participants will undergo a genetic comprehension questionnaire. Genetic information presents challenges to all participants within studies, but especially those with low and marginal genetic literacy. Low genetic comprehension may be a barrier for participants to understand the utility of the return of genetic results information, therefore, the investigatorswill measure genetic comprehension through the use of the questionnaire the Measure of Genetic Susceptibility Knowledge. This questionnaire will be administered orally to the study participants by the URB staff who will follow structured protocols. This questionnaire was created by selecting questions from previous questionnaires that measure genetic knowledge in the general population as well as creating comprehension questions from a previous questionnaire that used on this population called the Return of Results (Genetic) Questionnaire from IRB18-1331.

Participants in the intervention arms will also be given a questionnaire to measure any psychological stress due to receiving ROR. It is important to understand the psychological consequences for patients receiving genomic tests results in a variety of settings, therefore, the investigators will measure psychological stress through the use of the Feelings About genomiC Testing Results (FACToR) questionnaire, that has been designed to measure the psychological impact of receiving genomic test results in a wide range of conditions.

Additionally, participants identified the well water used as their primary source of drinking water at baseline in the HEALS cohort study, the investigators will follow-up on this question to have the most up to date information.

Potential risks and benefits: There is no more than minimal physical risk to participate in this study. The investigators are requesting to obtain urine samples and questionnaire data from all of the participants. While the study is no more than minimal physical risk/harm, the investigators will have numerous precautions to protect confidentiality.

Additionally, there may be some risk of stigma or stress to individuals in the intervention arm, who are identified as slow arsenic metabolizers, however, this is offset by the potential health benefit gained through the knowledge. According to the health belief model, if genetic risk information changes an individual's perceived susceptibility to arsenic toxicities, the likelihood to adopt health behaviors may change. Therefore, for the participants in this specific study who are at higher risk for arsenic toxicities due to having higher urine arsenic levels throughout the 15-20 years of follow-up data in the HEALS cohort, obtaining information regarding being a slower arsenic metabolizers may additionally motivate lifestyle modification if it increases an individual's risk perception, thereby offsetting the potential risk through this benefit. Furthermore, a subset of 200 participants in the HEALS study have previously been asked if they would like to receive their genetic information regarding arsenic metabolism efficiency, 100% of the participants questioned stated they would want this information.

Monitoring of Safety: This study involves no physical risks. The intervention is informational in nature, and occurs at a single point in time (i.e., the baseline visit). Should individuals want to further discuss the genetic information received with a health care professional, a contact number for a HEALS study physician will be provided to all participants. Furthermore, all HEALS participants can access free primary health care through the local HEALS clinic, should participants have any health concerns related the arsenic-related information received during participation in this study.

Procedure to obtain and record informed consent: For this present study, Uchicago Research Bangladesh (URB) study staff will work to identify patients who meet the inclusion and exclusion criteria from the established HEALS cohort study during which the URB staff will obtain informed consent.

Confidentiality: While the study is no more than minimal physical risk/harm, the investigators will have numerous precautions to protect confidentiality. The study does not involve the collection of identifiable information, and the URB study staff will assign a coded unique study ID to all participant data and samples. The investigators will ensure that all samples are coded, and all data will be protected, stored, and analyzed on secure password-protected servers in the Department of Public Health Studies (PHS) at the University of Chicago.

ELIGIBILITY:
For this present study, UChicago Research Bangladesh (URB) study staff will work to identify patients who meet our inclusion and exclusion criteria from our established HEALS cohort study during which the URB staff will obtain informed consent. The inclusion criteria for the study are:

* HEALS cohort members
* age 18-70
* consistently high urine arsenic levels (≥ 200 µg/g creatinine) based on 15-20 years of follow-up data
* existing data on genetic information regarding the AS3MT variants that classify them as being an inefficient or efficient arsenic metabolizer.

The exclusion criteria for this study would be HEALS members who are

* missing baseline urine samples
* missing the latest follow-up urine samples.

There will be a total of 300 subjects enrolled,100 for the intervention 1 group, 100 for the intervention 2 group and 100 for the control group.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
change in arsenic concentration in urine | six months
  Urine samples will be obtained by URB study staff at baseline (Time1 or initial contact) and Time2 (Six months after the onset of the intervention). Urine arsenic will be measured using Inductively Coupled Plasma Mass spectrometry (ICPMS) at the CACHET (The Chicago Center for Health and Environment) biomarkers core facility at UIC (University of Illinois at Chicago). The difference between arms in the change in arsenic from time 1 to time 2 will be assessing using regression-based statistical methods.

SECONDARY OUTCOMES:
Psychological stress | six months
  Participants in the intervention arms will also be given a questionnaire to measure any psychological stress due to receiving ROR. It is important to understand the psychological consequences for patients receiving genomic tests results in a variety of settings, therefore, we will measure psychological stress through the use of the Feelings About genomiC Testing Results (FACToR) questionnaire, that has been designed to measure the psychological impact of receiving genomic test results in a wide range of conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- UChicago Research Bangladesh, Dhaka, Dhaka-1230, Bangladesh

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-10-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT05072132/ICF_000.pdf